CLINICAL TRIAL: NCT03859856
Title: Ovarian Reserve in Patients With Type 1 Diabetes Mellitus
Brief Title: Ovarian Reserve in Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Aslan Cetin, Md, ObGYN, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2018.10.23
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-02

CONDITIONS: Type1 Diabetes Mellitus
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women with Type 1 diabetes mellitus: Reproductive age women diagnosed with type 1 diabetes mellitus
  Interventions: Other: hormone panel and ultrasonography
- women without Type 1 diabetes mellitus: Reproductive age women diagnosed with type 1 diabetes mellitus to serve as control
  Interventions: Other: hormone panel and ultrasonography

INTERVENTIONS:
Other: hormone panel and ultrasonography — Blood sampling on the 3rd day of menstrual cycle for the measurement of serum FSH, LH, E2 and AMH hormone levels and ultrasonography for antral follicle count and ovarian volume measurement will be done.

SUMMARY:
Type 1 diabetes mellitus is a common autoimmune disease. It affects women of all ages including reproductive years. Hyperglycemic condition in diabetes can cause organ damage. This study aims to measure serum hormones including FSH, LH, E2, AMH, ovarian volume and antral follicle count (indicators of ovarian reserve) in women with and without type 1 diabetes mellitus.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus is a common autoimmune disease. It affects women of all ages including reproductive years. It is showed that hyperglycemic state in diabetes results in organ damage like kidneys and eyes. Ovarian reserve is important for the reproductive period. The measurements of serum hormones including follicle stimulating hormone (FSH), luteinizing hormone (LH), estradiol (E2) and anti-mullerian hormone (AMH) will give us an idea about the ovarian reserve. The investigators aim is to measure ovarian reserve parameters in patients diagnosed with type 1 diabetes mellitus and to compare them to healthy controls. Serum FSH, LH, E2 and AMH will be measured on the 3rd day of the cycle. Antral follicle count and ovarian volume measurement will be done with ultrasonography. Ovarian reserve markers will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive age group women: 18-40 years
* Women diagnosed with type 1 diabetes (case group)
* Women without type 1 diabetes (control group)

Exclusion Criteria:

* Women with PCOS (polycystic ovary syndrome)
* history of ovarian surgery
* Body mass index (BMI) over 30

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be reproductive age women diagnosed with type 1 diabetes mellitus. The control population will be aged and BMI matched women without type 1 diabetes mellitus.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-11-25 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
E2, FSH, LH, AMH levels | during procedure
  E2, FSH, LH, AMH levels of blood samples will be measured
antral follicle count | during procedure
  antral follicles of ovaries will be counted with ultrasonography
ovarian volume | during procedure
  both ovaries will be measured in three dimensions with ultrasonography

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni SSTRH, Istanbul, Turkey (Türkiye)